CLINICAL TRIAL: NCT01328678
Title: A Pilot Study of Vitamin D in Subjects With Alopecia Areata
Brief Title: A Study of Vitamin D in Subjects With Alopecia Areata
Status: Completed | Type: Observational
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Wael Eid, MD, Avera McKennan Hospital & University Health Center
Other Study IDs: ARI-1270-Alopecia
Record Dates: First submitted 2011-01-06; First posted 2011-04-05 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2011-07

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata; Vitamin D; Parathyroid; Calcium
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Alopecia Areata: Individuals with Alopecia Areata (AA)

SUMMARY:
The objective of this study is to assess the parathyroid-vitamin D-calcium axis in subjects with alopecia areata. The hypothesis behind this study is that hypovitaminosis D might contribute to the pathogenesis of alopecia areata.

DETAILED DESCRIPTION:
Alopecia Areata (AA) is a T-Cell mediated, non-scarring, polygenic, autoimmune disease of the hair follicle. It has been reported to be associated with other autoimmune diseases, especially autoimmune thyroid disease and vitiligo. It is more common in females. Recently, vitamin D deficiency has been claimed to contribute to the pathogenesis of multiple autoimmune disease. There is a strong inverse correlation between the level of 25-hydroxyvitamin D levels and the autoimmune disease in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are at least 18 years old
* Subjects with newly diagnosed with alopecia areata

Exclusion Criteria:

* Subjects who take supplemental Vitamin D, by itself or as a part of a multivitamin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women in and around the Sioux Falls area
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Vitamin D levels will be reported in subjects and correlated with the calcium and parathyroid levels. | Initial clinic visit (day 1)
  This study consists of a single clinic visit. After subject has completed the informed consent process and meets eligibility criteria, a blood sample will be collected. Lab results from this one-time lab draw will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Wael Eid, MD, Principal Investigator — Avera McKennan Hospital & University Health Center
Locations (1):
- Avera Research Institute, Sioux Falls, South Dakota, United States